CLINICAL TRIAL: NCT03069586
Title: The Effect of Low Pressure Pneumoperitoneum and Pulmonary Recruitment Manoeuvre on Postoperative Pain After Laparoscopic Cholecystectomy
Brief Title: Effect Low Pressure Pneumoperitoneum and Pulmonary Recruitment on Postoperative Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: General Hospital Groeninge (Other)
Responsible Party: Principal Investigator, Casier Isabelle, Doctor, General Hospital Groeninge
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AZGS2014160
Record Dates: First submitted 2016-02-10; First posted 2017-03-03 (Actual); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Pneumoperitoneum; Recruitment; Postoperative Pain
MeSH Terms: conditions — Pneumoperitoneum; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low pressure pneumoperitoneum (Other): Surgery on low pressure pneumoperitoneum (8 - 10 mmHg).
  Interventions: Procedure: No pulmonary recruitment
- low pressure peritoneum and pulmonary recruitment (Active Comparator): Surgery on low pressure pneumoperitoneum (8 - 10 mmHg) and at the end of surgery a manual pulmonary recruitment manoeuver (2 x 5sec max 40cmH2O) will be done
  Interventions: Procedure: Pulmonary recruitment

INTERVENTIONS:
Procedure: Pulmonary recruitment — At the end of surgery a manual pulmonary recruitment (5 sec, max 40 cmH2O) is given to the patiënt
  Arms: low pressure peritoneum and pulmonary recruitment
Procedure: No pulmonary recruitment — At the end of surgery no intervention was completed
  Arms: Low pressure pneumoperitoneum

SUMMARY:
The investigators want to test the hypothesis that the addition of a recruitment manoeuvre to a low pressure pneumoperitoneum will lead to an additional reduction in postoperative pain. Therefore the investigators will conduct a prospective randomized controlled, single blind trial.

DETAILED DESCRIPTION:
Two groups:

1. A cholecystectomy at a low pressure pneumoperitoneum (8-10 mmHg)
2. A cholecystectomy at a lowpressure pneumoperitoneum (8-10mmhg) and at the end a pulmonary recruitment manoeuvre (5 sec at max 40 cmH2O).

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II

Exclusion Criteria:

* refusal to give consent
* cholecystitis
* BMI above 35
* intolerance to one of the pain medication
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-03 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
pain relief during the first 24 hours | 24hours
  VAS (0-10)

SECONDARY OUTCOMES:
Total analgesic use during the first 24 hours | 24hours
Length of hospital stay | 2 days
Recovery after 48 hours | 48 hours
  quality of recovery scale

CONTACTS AND LOCATIONS:
Locations (1):
- AZ groeninge, Kortrijk, Belgium

IPD SHARING:
Plan to Share IPD: No